CLINICAL TRIAL: NCT00428480
Title: Stroke Inpatient Rehabilitation Reinforcement of Walking Speed
Brief Title: Walking Study for Stroke Rehabilitation
Acronym: SIRROWS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: WORLD FEDERATION FOR NEUROREHABILITATION (Unknown); Mayo Clinic (Other); The Foundation Institute San Raffaele G. Giglio of Cefalù (Other); University of Vigo (Other); Morinomiya Hospital, Osaka, Japan (Unknown); Chonnam National University Hospital (Other); Asklepios Kliniken Hamburg GmbH (Other); Burke Rehabilitation Hospital (Other); Hacettepe University (Other); Department of Rehabilitation, University Hospital, Czech Republic (Other); Federal Medical Center, Abeokuta, Nigeria (Unknown); Ankara University (Other); Institute for Clinical Research (Other); University of Chicago (Other); Helen Hayes Hospital (Other); Gazi University (Other); All India Institute of Medical Sciences (Other); Shirley Ryan AbilityLab (Other); St. Luke's Hospital, Pennsylvania (Other); Hochzirl Hospital (Other); Father Muller Medical College (Other); Kernan Hospital, Baltimore (Unknown); IRCCS San Camillo, Venezia, Italy (Other); Kessler Foundation (Other); Vanderbilt Stallworth Rehabilitation Hospital, TN (Unknown); Rehabilitation Hospital of Rhode Island, RI (Unknown); St. Mauritius Therapieklinik, Dusseldort, Germany (Unknown)
Responsible Party: Dr. Bruce Dobkin, University of California Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCLA-06-07-104-01
Record Dates: First submitted 2007-01-29; First posted 2007-01-30 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2009-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Daily reinforcement of walking speed
  Interventions: Behavioral: Daily reinforcement of walking speed (DRS)
- 2 (Active Comparator): No reinforcement of walking speed
  Interventions: Behavioral: No reinforcement of walking speed (NRS)

INTERVENTIONS:
Behavioral: Daily reinforcement of walking speed (DRS) — Inpatients are encouraged to walk faster and given feedback on their walking speed during a daily 10-meter walk as part of their usual physical therapy.
  Other Names: DRS
  Arms: 1
Behavioral: No reinforcement of walking speed (NRS) — Inpatients complete a 10-meter walk as part of their daily physical therapy but are not given any encouragement to walk faster or feedback on their walking speed.
  Other Names: NRS
  Arms: 2

SUMMARY:
The primary purpose of this study is to determine the effects of reinforcement of walking speed on recovery of walking speed over the course of inpatient rehabilitation for people after stroke. The study will also examine the relationship between short distance walking speed and walking distance over a fixed time.

DETAILED DESCRIPTION:
This study is a single-blind, randomized, multi-center trial design. People who are admitted post-stroke for inpatient rehabilitation will be examined for eligibility by the treating physician. Subjects who satisfy the selection criteria and who agree to participate will be randomized to either the experimental group or the control group.

Intervention

All subjects will receive usual therapy during their inpatient rehabilitation stay.

Subjects in the experimental group (Daily Reinforcement of Speed or DRS group) will receive encouragement to walk faster with feedback on their performance every day for the duration of their inpatient stay. During one of the daily therapy sessions (preferably morning), the experimental subjects will be encouraged by their physical therapist to walk at least 10 m (25 feet) along a straight hallway. Subjects in the experimental group will be timed with a stopwatch by their treating physical therapist each day during the 10-meter walking task. If a subject is not able to walk 10 meters, then a shorter distance is used until the 10-meter distance can be achieved (if possible). Before starting the timed walk, the therapist will remind the subject to "walk as fast as safely possible" and to try to walk the distance "a few seconds faster than what you were able to do in the past few days". The therapist can provide the assistance of another person and use aids, and whatever is needed for safety. The timed test should be stopped or not performed on any one day if this is best for patient care. The subject's safety must not be compromised. At the end of the timed walk, the therapist will provide the results for that day in a positive tone, such as "Very good! You walked that in xx seconds". Then, (a) 'This is better by x seconds', or (b) 'This shows you are holding your own', or (c) 'I believe that you will soon be able to walk a bit faster with a better walking pattern'."

Subjects who are randomized to the control group (No Reinforcement of Speed or NRS group) will not be timed during a daily 10-meter walk, nor specifically encouraged to walk faster each day.

Outcome measures

The primary outcome measure is walking speed, measured with a stopwatch over 15.2 m (50 feet).3 A blinded evaluator (i.e. a physical therapist or other trained person who is not involved in the subject's treatment and does not work on the inpatient unit) will conduct all assessments. The treating physical therapist will assist the subject during the gait speed assessments as necessary. The subject will employ his or her usual assistive devices for that stage of recovery.

The gait speed assessment will be conducted on a flat tiled surface along a walkway that is not within sight of other patients. A chair will be placed at either end of the 15 m straight walkway. The subject starts approximately 3 steps behind the start line to allow for acceleration. The blinded assessor instructs the subject to "walk as fast as you safely can until I tell you to stop. If you have to sit or rest, tell me." When the subject's lead toe crosses the line, timing begins. When the lead toe crosses the 15.2-meter (finish) line, timing stop. The subject is told to stop walking once both feet cross the line. This ensures that the subject does not decelerate until he or she has traversed the full 15.2 meters. Data is recorded as time in seconds.

At entry to the study, it is anticipated that some subjects may not be able to walk continuously for 15 meters. In these cases, a timed 5-meter walk can be substituted at study entry and designated so on the data entry form, and if still necessary, at discharge. If a subject at study entry cannot walk 5 meters without stopping to rest or needs maximal assistance, the test is marked "unable" on the data recording sheet.

Gait speed measurements will be collected by the blinded evaluator at study entry (if possible), at 1, 2, 4, 6, and 8 weeks after entry if still an inpatient, within one day of inpatient discharge, and, if possible, 3 months and 6 months after study entry. The Functional Ambulation Classification Index will be completed by the blinded evaluator after each gait speed assessment. Thus, a FAC score will be recorded at the same time points as each gait speed evaluation.

The secondary outcome measure is distance walked in 3 minutes. The subject will be instructed by the blinded assessor to walk as many laps of the walkway as possible in 3 minutes. A straight 25-meter walkway will be used. The patient turns at each end and continues walking for the 3 minutes. The distance covered in 3 minutes is measured in meters. The subject may halt to rest at any time and continue walking when ready. If the subject must sit down to rest, the test is discontinued and the time and distance are recorded. The 3-minute walking test will be conducted at up to 4 time points: 4 weeks after entry if still an inpatient, within 2 days of inpatient discharge, 3 months post study entry, and 6 months post study entry. If the evaluator believes that the test was not an accurate reflection of the walking distance (some interruption occurred or the subject stopped when distracted), the test can be repeated and the best distance recorded.

The blinded observer should find an isolated and convenient place to perform the tests. Before the trial begins, the observer should practice the timed walking speed and distance test with 3 hemiparetic inpatients and their therapists for 4 repeated tests within 1-2 days to try to obtain reproducible data. The walking speeds and distances should not differ by more than 10%.

Descriptive data and further assessments

Each subject will have data recorded by site and randomization number, not by name, birth date or other identifying characteristics. In addition to the results from the gait speed and walking distance assessments (collected and entered by the blinded evaluator), basic descriptive information for each subject will also be collected in order to adequately characterize the study population. This information will be obtained by the study physician or designated person from the medical record and from interview with the subject or family. The following information will be collected for each subject: age, gender, handedness; dates of stroke onset, admission for rehabilitation, entry into the trial, and discharge from in patient care; and (selected from a list) type of stroke, general location of stroke, and side of hemiparesis. Severity of stroke at the time of entry into the study will be characterized using the National Institutes of Health Stroke Scale,4-5 the modified Rankin Scale, and the Functional Ambulation Classification Index, which are well accepted measures. The investigators will also ask subjects to record the number of falls they had from discharge to 3 months and from 3 months to 6 months after entry using a calendar that they will bring with them to each follow-up.

Data entry

All data entry will be via a web-based system. The blinded observer will enter all walking-related data and will be given a password to access the data entry site that differs from the password and access by the study physician.

Data analysis

For an anticipated effect size of 0.4, a conservative estimate using a two-tailed alpha of 0.01 and power of 0.9, we will need a sample size of 150 subjects in each group. An ideal sample size for this varied population and for the primary and secondary outcomes will be 250 subjects in each arm to allow for dropouts and to gather enough subjects who are also tested at 3 and 6 months study entry. This would make the trial the largest prospective neurorehabilitation study ever attempted.

ELIGIBILITY:
Inclusion Criteria:

* 35 years or older
* suffered a stroke from any cause that is unlikely to progress or recur within 2 years of onset (thrombotic infarct, cardioembolus, intracerebral hemorrhage)
* unilateral hemiparesis with strength of the proximal leg muscles ≤4/5
* able to follow simple instructions and understand verbal reinforcement about walking speed
* able to take 5 steps with not more than the assistance of one person

Exclusion Criteria:

* premorbid walking difficulty in the community, such as a prior stroke with residual impairment, arthritis with pain on stepping, dyspnea or angina on modest exertion, limited walking endurance due to cardiopulmonary or other disease
* history of dementia
* current medical disease that will limit physical therapy at the time of randomization, such as critical illness myopathy/neuropathy, serious infection, thrombophlebitis, orthostatic hypertension, decubitus ulcer, congestive heart failure, chronic obstructive lung disease, organ transplantation, recent surgery (including coronary bypass), or pain with weigh bearing

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2007-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Gait speed | Admission, 2 weeks, 4 weeks, 6 weeks, 8 weeks, discharge, 3 months, 6 months

SECONDARY OUTCOMES:
Distance walked in 3 minutes | 4 weeks, discharge, 3 months, 6 months
Functional Ambulation Classification (FAC) | Admission, 2 weeks, 4 weeks, 6 weeks, 8 weeks, discharge, 3 months, 6 months
Number of falls post inpatient rehabilitation | 3 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bruce H Dobkin, MD, Principal Investigator — University of California, Los Angeles
Locations (24):
- United States (11):
  - University of California Los Angeles, Los Angeles, California
  - The Rehabilitation Institute of Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Kernan Hospital, Baltimore, Maryland
  - St. Luke's and Whiteside Institute for Clinical Research, Duluth, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Kessler Medical Rehabilitation Research and Education Corporation, West Orange, New Jersey
  - Burke Rehabilitation Hospital, White Plains, New York
  - St. Luke's Hospital, Bethlehem, Pennsylvania
  - Rehabilitation Hospital of Rhode Island, North Smithfield, Rhode Island
  - Vanderbilt Stallworth Rehabilitation Hospital, Nashville, Tennessee
- Hospital Hochzirl, Zirl, Austria
- St. Mauritius Therapieklinik, Düsseldorf, Germany
- India (2):
  - Father Muller Medical College, Mangalore, Karnataka
  - All India Institute of Medical Sciences, New Dehli
- Italy (3):
  - Fondazione Instituto San Raffaele-Giglio, Cefalù
  - University of Salute, San Raffaele Hospital, Milan
  - I.R.C.C.S San Camillo, Venezia
- Morinomia Hospital, Osaka, Japan
- Federal Medical Center, Abeokuta, Nigeria
- Chonnam National Medical School & Hospital, Gwangju, South Korea
- University Hospital of Vigo, Vigo, Spain
- Turkey (Türkiye) (2):
  - Ankara University Faculty of Medicine, Ankara
  - Gazi University Faculty of Medicine, Ankara